CLINICAL TRIAL: NCT01670136
Title: Pharmacokinetics of Sildenafil in Premature Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-1646; HHSN27500014 (Other Grant/Funding Number: NICHD)
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Persistent Pulmonary Hypertension of the Newborn
Keywords: sildenafil; preterm infants; persistent pulmonary hypertension of the newborn
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sildenafil, standard of care (No Intervention): Infants receiving sildenafil as standard of care
- sildenafil administered for study (Other): 1 dose of sildenafil administered for study
  Interventions: Drug: 1 dose of sildenafil

INTERVENTIONS:
Drug: 1 dose of sildenafil — A single IV dose of sildenafil will be administered over 90 minutes with no greater than a 15-minute flush. Final dose to be determined based on at least the first 4 participants enrolled in Cohort 1; final dose expected to be a single dose between 0.25 and 0.5 mg/kg.
  Other Names: Revatio; Viagra
  Arms: sildenafil administered for study

SUMMARY:
The purpose of this study is to learn more about the safety and dosing of sildenafil in infants.

DETAILED DESCRIPTION:
Pharmacokinetics and safety of sildenafil will be studied in preterm infants who are receiving sildenafil per standard of care or 1 dose prescribed for the study.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

* Gestational age 28 weeks or less receiving sildenafil as standard of care < 365 postnatal days

Cohort 2:

* Gestational age 28 weeks or less
* 7-28 postnatal days of age
* Mechanical ventilation or nasal continuous positive airway pressure (NCPAP) or high-flow nasal cannula
* Intravenous line in place

Exclusion Criteria:

Cohort 1:

* Any condition that would make the participant, in the opinion of the investigator, unsuitable for the study

Cohort 2:

* Previous exposure to sildenafil within 7 days prior to enrollment
* Any condition that would make the participant, in the opinion of the investigator, unsuitable for the study
* History of allergic reactions to sildenafil
* AST > ULN or ALT > 3x ULN
* Currently on a vasopressor for hypotension
* Known sickle cell disease

Max Age: 364 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2013-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve 0-24 hours for sildenafil | IV study dose 0-15 min,1-2,3-4,12-14,24-30,48-56hr after flush.Clinical care: IV <0.5hr before dose <15 min & 3-4hr after flush <0.5hr before next dose. Enteral <0.5hr before dose, 1-2 & 3-4hr after dose, <0.5hr before next dose. 22-26hr after last dose
Peak plasma concentration of sildenafil | IV study dose 0-15 min,1-2,3-4,12-14,24-30,48-56hr after flush.Clinical care: IV <0.5hr before dose <15 min & 3-4hr after flush <0.5hr before next dose. Enteral <0.5hr before dose, 1-2 & 3-4hr after dose, <0.5hr before next dose. 22-26hr after last dose
Clearance of sildenafil | IV study dose 0-15 min,1-2,3-4,12-14,24-30,48-56hr after flush.Clinical care: IV <0.5hr before dose <15 min & 3-4hr after flush <0.5hr before next dose. Enteral <0.5hr before dose, 1-2 & 3-4hr after dose, <0.5hr before next dose. 22-26hr after last dose
Volume of distribution at steady state | IV study dose 0-15 min,1-2,3-4,12-14,24-30,48-56hr after flush.Clinical care: IV <0.5hr before dose <15 min & 3-4hr after flush <0.5hr before next dose. Enteral <0.5hr before dose, 1-2 & 3-4hr after dose, <0.5hr before next dose. 22-26hr after last dose
Half life of sildenafil | IV study dose 0-15 min,1-2,3-4,12-14,24-30,48-56hr after flush.Clinical care: IV <0.5hr before dose <15 min & 3-4hr after flush <0.5hr before next dose. Enteral <0.5hr before dose, 1-2 & 3-4hr after dose, <0.5hr before next dose. 22-26hr after last dose

SECONDARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability. | From the time of the first dose to 3 days after the last dose; serious adverse events will be collected from the first dose of sildenafil to 7 days after the last dose of sildenafil
Correlation between serum and dried blood spot samples | 1-7 days
Evaluate P450 single nucleotide polymorphisms (SNPs) | 2-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Laughon, MD, MPH, Principal Investigator — University of North Carolina
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Riley Hospital, Indianapolis, Indiana
  - Kosair Pediatric Research Unit, Louisville, Kentucky
  - Albany Medical Center, Albany, New York
  - Kings County Hospital Center/SUNY Downstate Medical Center, Brooklyn, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jackson W, Gonzalez D, Smith PB, Ambalavanan N, Atz AM, Sokol GM, Hornik CD, Stewart D, Mundakel G, Poindexter BB, Ahlfeld SK, Mills M, Cohen-Wolkowiez M, Martz K, Hornik CP, Laughon MM; Best Pharmaceuticals for Children Act-Pediatric Trials Network Steering Committee. Safety of sildenafil in extremely premature infants: a phase I trial. J Perinatol. 2022 Jan;42(1):31-36. doi: 10.1038/s41372-021-01261-w. Epub 2021 Nov 5. PMID 34741102